CLINICAL TRIAL: NCT07250334
Title: Prospective Phase I/II Study Evaluating the Safety and Efficacy of Preoperative Carbon Ion Radiotherapy in Patients With Soft Tissue Sarcoma : The SARCOMA-01 Trial by the Severance sARCOma Multidisciplinary Team
Acronym: SARCOMA-01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-1025
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIRT Group (Experimental): Phase I (Dose-Escalation) Participants in the Phase I cohort will receive preoperative CIRT using a dose-escalation design to identify an optimal tolerated dose. Three dose levels are evaluated-32.0, 34.0, and 36.0 GyE/8 fractions-delivered in 2 weeks (4 fr/week). Surgical resection is performed 6-8 weeks after CIRT, followed by postoperative evaluation of wound healing, toxicity, and surgical outcomes.
  Phase II (Feasibility and Safety Evaluation) All enrolled patients will receive preoperative CIRT at the optimal dose determined in Phase I. The regimen consists of 8 fractions (4 fr/week), followed by surgical resection 6-8 weeks later. Postoperative assessments focus on feasibility and safety, particularly grade 3-5 wound complications within 120 days after surgery. Secondary analyses include pathological response, R0 resection rate, local control, survival, and quality of life. Participants are followed for at least 12 months to assess long-term safety and efficacy.
  Interventions: Radiation: Carbon-Ion Radiotherapy (CIRT)

INTERVENTIONS:
Radiation: Carbon-Ion Radiotherapy (CIRT) — Participants receive preoperative CIRT as the investigational intervention, delivered in 8 fractions, once daily, four times per week. In Phase I, three dose levels (DL1: 32.0 GyE, DL2: 34.0 GyE, DL3: 36.0 GyE) are evaluated using a 3+3 dose-escalation design to determine the recommended Phase II dose (RP2D). Three patients are initially enrolled per dose level, expanded to six if dose-limiting toxicities occur. In Phase II, all participants receive CIRT at the RP2D following a Simon's two-stage design (Stage I: 20 patients; Stage II: 22 additional if criteria met). Treatment uses fixed-beam or rotating gantry techniques. Post-treatment imaging (CT or MRI) is performed 4-6 weeks after CIRT, followed by surgical resection 6-8 weeks post-radiotherapy. All participants are followed for at least 12 months after surgery to assess postoperative wound complications, treatment completion, and overall outcomes.

SUMMARY:
"This prospective, single-institution Phase I/II clinical trial investigates the safety, feasibility, and preliminary efficacy of preoperative carbon-ion radiotherapy (CIRT) for patients with resectable soft tissue sarcoma. Given the radioresistant nature of sarcomas and the limitations of photon-based preoperative radiotherapy-particularly high wound complication rates-CIRT is expected to enhance local tumor control while minimizing treatment-related toxicity and surgical morbidity.

The trial consists of an initial dose-escalation phase (phase 1) to identify an optimal and tolerable dose level, followed by an expansion phase (phase 2) assessing the feasibility of completing both CIRT and surgery without major wound complications. CIRT is delivered in eight fractions over two weeks, with surgery planned 6-8 weeks after radiotherapy.

Primary endpoints include the incidence of grade 3-5 post-operative wound complications within 120 days and overall treatment completion. Secondary endpoints include pathological response, surgical outcomes, local control, progression-free survival, overall survival, and patient-reported quality of life. All participants will be followed for at least 12 months postoperatively to evaluate safety and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older.
* Histologically confirmed soft tissue sarcoma deemed suitable for curative resection.
* Determined by the Yonsei Cancer Center sarcoma multidisciplinary team that preoperative carbon-ion radiotherapy followed by surgery is appropriate, considering tumor histologic subtype, size, and location.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 or Karnofsky Performance Status (KPS) ≥ 70.
* Adequate organ function (including hematologic, hepatic, and renal function) suitable for radiotherapy and surgery.
* Voluntarily provided written informed consent.

Exclusion Criteria:

* Presence of distant metastases.
* Inability to plan carbon-ion radiotherapy due to metallic implants or other factors at the tumor site.
* History of prior radiotherapy to the same anatomical region.
* Presence of other serious medical conditions or active infections that, in the investigator's judgment, could interfere with study participation.
* Presence of active implanted electronic devices (e.g., pacemaker or defibrillator) without established safety for carbon-ion radiotherapy.
* Pregnant or breastfeeding women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence of Dose-Limiting Toxicities (DLTs) | From initiation of CIRT to 30 days after surgery
  To evaluate the safety and tolerability of preoperative CIRT and identify the optimal tolerated dose level. DLTs are defined as grade ≥3 toxicities, including severe wound complications, prolonged hospitalization, or significant treatment delay, assessed according to CTCAE version 5.0.
Phase II: Proportion of Patients Completing Both CIRT and Surgery Without Grade 3-5 Postoperative Wound Complications or Serious Adverse Events | From initiation of CIRT to 120 days after surgery
  To determine the clinical feasibility and safety of completing preoperative CIRT followed by surgical resection without major wound-healing complications or treatment-related serious adverse events (SAEs). The endpoint represents the proportion of patients achieving treatment completion without grade 3-5 wound complications or other SAEs within 120 days postoperatively.

SECONDARY OUTCOMES:
Incidence of Acute Treatment-Related Toxicities | From initiation of CIRT to 30 days after surgery
  To record and grade all acute adverse events associated with preoperative carbon-ion radiotherapy using CTCAE v5.0 criteria to characterize the overall safety profile at each dose level.
Surgery Feasibility and Completion Rate | From completion of CIRT to 30 days after surgery
  To assess the proportion of participants who successfully undergo and complete surgical resection following preoperative CIRT without protocol deviation or treatment interruption.
Pathological Tumor Response Rate | At surgical specimen evaluation (6-8 weeks after CIRT)
  To determine the rate of pathological tumor regression or necrosis in resected specimens following preoperative CIRT, based on standardized histologic grading criteria.
R0 Resection Rate | At surgery (6-8 weeks after CIRT)
  To evaluate the proportion of patients achieving microscopically margin-negative (R0) resection after preoperative CIRT, reflecting its impact on surgical resectability.
Local Control and Progression-Free Survival | From date of surgery to 12 months postoperatively
  To estimate 1-year local control and progression-free survival using Kaplan-Meier analysis as measures of preliminary efficacy.
Overall Survival | From initiation of CIRT to 12 months postoperatively
  To evaluate 12-month overall survival as an exploratory efficacy endpoint of preoperative CIRT.
Quality of Life (EORTC QLQ-C30) | Baseline, post-CIRT, and 3, 6, and 12 months after surgery
  To assess longitudinal changes in patient-reported quality of life using the EORTC QLQ-C30 questionnaire throughout treatment and follow-up.
Body Composition Change (InBody Analysis) : Skeletal-Muscle Mass Change | Baseline, post-CIRT, and 3, 6, and 12 months after surgery
  Unit of Measure: kg
Body Composition Change (InBody Analysis) :Body-Fat Composition Change | Baseline, post-CIRT, and 3, 6, and 12 months after surgery
  Body-Fat Composition Change

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center, Yonsei University College of Medicine, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No